CLINICAL TRIAL: NCT04583514
Title: Testing the Adipose Expandability Hypothesis in Vivo During Overfeeding
Acronym: EAT 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ursula White, Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PBRC 2019-051; R01DK121944 (NIH)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Overweight and Obesity; Metabolic Syndrome
Keywords: Overweight; Adipose tissue; Subcutaneous abdominal; Subcutaneous femoral; Adipocyte; Adipose turnover; Adipose kinetics; Adipogenesis; Ectopic fat; Insulin sensitivity; Deuterium
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): The control group will be expected to maintain their weight within 1 kg of baseline weight throughout the duration of the study.
  Interventions: Behavioral: Control
- Overfeeding (Experimental): The overfeeding group will be subjected to a similar relative change in energy intake, in which their dietary intake will be 30% more kcal/d than needed for weight maintenance.
  Interventions: Behavioral: Overfeeding

INTERVENTIONS:
Behavioral: Control — Weight-stable Control group
  Arms: Control
Behavioral: Overfeeding — 30% Overfeeding group
  Arms: Overfeeding

SUMMARY:
Adipose, or fat, tissue is a plastic organ that retains the ability to expand and store excess calories during positive energy balance in humans. The capacity of subcutaneous (subQ) adipose tissue to expand and remodel is an important determinant of obesity-related health complications, and impaired expansion of subQ fat tissue is thought to contribute to the risk of diseases such as the Metabolic Syndrome (MetS) and type 2 diabetes mellitus (T2D). The objectives of the study are to evaluate the changes and mechanisms of (subQ) adipose tissue expandability that occur as a result of short-term weight gain and to investigate the effects on cardio-metabolic health outcomes. Findings from this study will provide new insight into the dynamics of adipose expansion and remodeling during changes in energy balance and how this may impact future fat tissue function and metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Men and pre-menopausal women
* 18-42 years of age
* BMI 23-35 kg/m2 (± 0.5 will be accepted)
* Are willing to drink deuterium-labeled water (2H2O) for 8 weeks
* Are willing to be randomized to either a CTL or 30% OF group
* For women, if not using pharmaceutical (hormonal) contraception (i.e. birth control pills, vaginal ring, injections, or implant), must agree to use either a double barrier method as a form of birth control to prevent pregnancy (i.e. male condom with spermicide, with or without cervical cap or diaphragm); use implants or intrauterine contraceptive devices; have a tubal ligation (surgically sterile); practice abstinence; or be in an established relationship with a vasectomized or same sex partner during the entire duration of the study
* Must be willing to adhere to all study procedures, including attendance at all study visits
* If enrolled, agree to maintain the same level of physical activity throughout the duration of the study
* Must be willing to have blood stored for future research

Exclusion Criteria:

* Unstable weight in the last 3 months (± ~5% weight change)
* Diagnosis of Type 1 or 2 diabetes or a fasting blood glucose > 110 mg/dL
* Average screening blood pressure > 140/90 mmHg
* Diagnosis of major organ disease (e.g. heart, kidney, lung, thyroid, liver disease) or abnormal liver enzymes that are, in the opinion of the MI, clinically significant and represent a problem for study inclusion.
* Self-reported positive test for human immunodeficiency virus, hepatitis B or hepatitis C
* Any current or previous eating disorders
* Chronic use of systemic glucocorticoids (steroids), systemic adrenergic-stimulating agents, beta-blockers, antipsychotic medications, thiazolidinediones and other medications that may cause clinically significant weight gain or loss)
* Chronic use of prescription weight loss medications or over the counter weight loss medications which, in the opinion of the MI, will impact the study
* Chronic use of anti-depressant medications for less than 3 months
* Chronic smokers or users of tobacco products who cannot abstain for the duration of the inpatient visits
* Previous bariatric or other surgeries for obesity
* Had cancer in the last 5 years (some skin cancers acceptable)
* Pregnancy, breastfeeding, or planned pregnancy for the upcoming 6 months
* Partial or full hysterectomy
* PCOS
* Diagnosed psychotic conditions.

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue expansion and remodeling -- in vivo adipocyte formation | 8 weeks
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is enriched into the DNA of newly synthesized cells. The primary outcome is to assess changes in new adipocyte formation in vivo and other mechanisms of adipose expansion and remodeling in response to 30% overfeeding (OF group) relative to the weight-stable CTL group.

SECONDARY OUTCOMES:
Adipose tissue expansion and remodeling -- in vivo triglyceride synthesis | 8 weeks
  Following the consumption of deuterium-labeled water (2H2O; heavy water), adipose tissue biopsies from the subcutaneous abdominal and femoral depots will be collected. The 2H from the heavy water is incorporated into the glycerol component of the adipose, providing a measure of new triglyceride synthesis. A secondary outcome is to assess changes in triglyceride synthesis in vivo and other mechanisms of adipose expansion and remodeling in response to 30% overfeeding (OF group) relative to the weight-stable CTL group.
Cardiometabolic health outcomes | 8 weeks
  A secondary outcome is to investigate the correlation between mechanisms of adipose tissue expansion and remodeling with changes in metabolic health outcomes (i.e. abdominal adiposity; insulin sensitivity; ectopic lipid) in response to 30% OF relative to the CTL group.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula White, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States